CLINICAL TRIAL: NCT04483583
Title: Tailoring P2Y12 Inhibiting Therapy in Patients Requiring Oral Anticoagulation After Undergoing Percutaneous Coronary Intervention:The Switching Anti-Platelet and Anti-Coagulant Therapy (SWAP-AC) - 2 Study
Brief Title: Tailoring P2Y12 Inhibiting Therapy in Patients Requiring Oral Anticoagulation After PCI
Acronym: SWAP-AC-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202001360
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; dual antiplatelet therapy; oral anticoagulant
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ABCD-GENE >10 - Clopidogrel (Active Comparator): Patients with an ABCD-GENE>10 score will be randomized in a 1:1 fashion to ticagrelor (60 mg/bid) or clopidogrel (75 mg/qd). Treatment will be maintained for 30 days.
  Interventions: Drug: Clopidogrel
- ABCD-GENE >10 - Ticagrelor (Experimental): Patients with an ABCD-GENE>10 score will be randomized in a 1:1 fashion to ticagrelor (60 mg/bid) or clopidogrel (75 mg/qd). Treatment will be maintained for 30 days.
  Interventions: Drug: Ticagrelor 60mg
- ABCD-GENE <10 - Clopidogrel (Active Comparator): Patients with an ABCD-GENE<10 will be treated with clopidogrel (75 mg/qd) for 30 days.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor 60mg — Patients will be administered a 180 mg loading dose followed by a 60 mg bid for the duration of the study.
  Other Names: brilinta
  Arms: ABCD-GENE >10 - Ticagrelor
Drug: Clopidogrel — Patients will be administered a 600 mg loading dose followed by a 75 mg daily for the duration of the study.
  Other Names: plavix
  Arms: ABCD-GENE <10 - Clopidogrel; ABCD-GENE >10 - Clopidogrel

SUMMARY:
Clopidogrel is the P2Y12 inhibitor of choice in PCI patients requiring OAC. However, concerns have been raised based on the notion that a considerable number of patients may have inadequate response to clopidogrel. Although practice recommendations indicate that the use of potent P2Y12 inhibitors (i.e., ticagrelor) may be considered in patients at increased thrombotic risk, they do not recommend routine testing to identify patients with poor response to clopidogrel. The aim of this study is to assess the pharmacodynamic effects of different P2Y12 inhibiting therapy (clopidogrel vs ticagrelor) in patients at high risk for high platelet reactivity identified according to the ABCD-GENE score in PCI treated patients also requiring OAC. Up to a total of up to 63 patients are planned to be prospectively enrolled in this investigation which will entail a series of comprehensive pharmacodynamic assessments to reach the study aim.

DETAILED DESCRIPTION:
The combination of aspirin plus a P2Y12 receptor inhibitor, also known as dual antiplatelet therapy (DAPT), is the cornerstone of treatment for patients with coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI). However, a considerable number of patients undergoing PCI also have an indication to be on treatment with an oral anticoagulant (OAC). It is estimated that 10-15% of PCI patients also have an indication to be on OAC, raising concerns on their optimal antithrombotic treatment regimen. Studies have consistently shown dropping aspirin and maintaining a P2Y12 inhibitor and OAC to be associated with reduces bleeding without any significant increase in ischemic events. Accordingly, current practice recommendations is to limit the use of aspirin to the peri-PCI period and maintain dual therapy with a P2Y12 inhibitor and an OAC. Clopidogrel is the P2Y12 inhibitor of choice in PCI patients requiring OAC. However, concerns have been raised based on the notion that a considerable number of patients may have inadequate response to clopidogrel, also known as high platelet reactivity (HPR) status, and thus be at risk for thrombotic complications. Although practice recommendations indicate that the use of potent P2Y12 inhibitors (i.e., ticagrelor) may be considered in patients at increased thrombotic risk, they do not recommend routine testing to identify patients with HPR status. Nevertheless, consensus recommendations do indicate that the selective use of tests to define HPR status is a reasonable option in selected cases such as PCI patients requiring OAC. The aim of this study is to assess the pharmacodynamic effects of different P2Y12 inhibiting therapy (clopidogrel vs ticagrelor) in patients at high risk for HPR identified according to the ABCD-GENE score in PCI treated patients also requiring OAC. Up to a total of up to 63 patients are planned to be prospectively enrolled in this investigation which will entail a series of comprehensive pharmacodynamic assessments to reach the study aim.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Willing and able to provide written informed consent
* Undergone successful PCI and treated with DAPT (aspirin plus a P2Y12 inhibitor) per standard of care
* On treatment with a novel oral anticoagulant (apixaban, dabigatran, edoxaban, or rivaroxaban) for any indication (dosing regimen will be according to standard of care and at the discretion of the treating physician)

Exclusion criteria:

* Any active bleeding or history of major bleeding
* Ischemic Stroke within 1 month
* Any history of hemorrhagic stroke, or intracranial hemorrhage
* Known non-cardiovascular disease that is associated with poor prognosis (e.g., metastatic cancer) or that increases the risk of an adverse reaction to study interventions.
* End-stage renal disease on hemodialysis
* Known severe liver dysfunction or any known hepatic disease associated with coagulopathy
* History of hypersensitivity or known contraindication to clopidogrel or ticagrelor.
* Systemic treatment with strong inhibitors of both CYP 3A4 and p-glycoprotein (e.g., systemic azole antimycotics, such as ketoconazole, and human immunodeficiency virus [HIV]-protease inhibitors, such as ritonavir), or strong inducers of CYP 3A4, i.e.

rifampicin, rifabutin, phenobarbital, phenytoin, and carbamazepine

* Subjects who are pregnant, breastfeeding, or are of childbearing potential, and sexually active and not practicing an effective method of birth control (e.g. surgically sterile, prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization)
* Concomitant participation in another study with investigational drug
* Hemoglobin ≤9 mg/dL
* Platelet count <80x106/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortega-Paz L, Bor W, Franchi F, van den Broek WWA, Rollini F, Giordano S, Galli M, Been L, Ghanem G, Shalhoub A, Garabedian H, Al Saleh T, Uzunoglu E, Zhou X, Rivas A, Pineda AM, Suryadevara S, Soffer D, Mahowald MK, Choi CY, Zenni MM, Phoenix F, Ajjan RA, Ten Berg JM, Angiolillo DJ. P2Y12 Inhibition in Patients Requiring Oral Anticoagulation After Percutaneous Coronary Intervention: The SWAP-AC-2 Study. JACC Cardiovasc Interv. 2024 Jun 10;17(11):1356-1370. doi: 10.1016/j.jcin.2024.03.027. Epub 2024 Apr 7. PMID 38597172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no wash out or run-in periods.
Period: Overall Study
Arm/Group | ABCD-GENE >10 - Clopidogrel | ABCD-GENE >10 - Ticagrelor | ABCD-GENE <10 - Clopidogrel
Started | 20 | 19 | 42
Completed | 20 | 14 | 35
Not Completed | 0 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCD-GENE >10 - Clopidogrel | ABCD-GENE >10 - Ticagrelor | ABCD-GENE <10 - Clopidogrel | Total
Number analyzed (Participants) | 20 | 19 | 42 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.6) | 74.2 (10.2) | 70.1 (7.7) | 72 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: count (%)
  Participants
    Female | 8 | 8 | 5 | 21
    Male | 12 | 11 | 37 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: count (%)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 2 | 1 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 4 | 3 | 10
    White | 15 | 14 | 39 | 68
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
PCI indication [Count of Participants; unit: Participants]
  Stable Ischemic Heart Disease | 13 | 9 | 24 | 46
  Unstable angina | 4 | 3 | 7 | 14
  Non-ST-Segment Elevation Myocardial Infarction | 3 | 4 | 7 | 14
  ST-elevation myocardial infarction | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured as PRU
Description: The primary end point of our study will be levels of platelet reactivity, measured as P2Y12 reaction units (PRU) using the VerifyNow system of ticagrelor versus clopidogrel in patients with an ABCD-Gene score ≥10. A PRU >208 suggests high platelet reactivity, while <85 may indicate increased bleeding risk.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: PRU
Arm/Group | ABCD-GENE >10 - Clopidogrel | ABCD-GENE >10 - Ticagrelor | ABCD-GENE <10 - Clopidogrel
Number analyzed (Participants) | 20 | 14 | 35
PRU | 154.5 [77.5 to 183.5] | 23 [3 to 46] | 104 [35 to 167]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Our definition of adverse event and/or serious adverse event did not differ from the one of clinicaltrials.gov
Arm/Group | ABCD-GENE >10 - Clopidogrel | ABCD-GENE >10 - Ticagrelor | ABCD-GENE <10 - Clopidogrel
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/42
Other Adverse Events (participants affected / at risk) | 0/20 | 7/20 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABCD-GENE >10 - Clopidogrel (N=20) | ABCD-GENE >10 - Ticagrelor (N=20) | ABCD-GENE <10 - Clopidogrel (N=42)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABCD-GENE >10 - Clopidogrel (N=20) | ABCD-GENE >10 - Ticagrelor (N=20) | ABCD-GENE <10 - Clopidogrel (N=42)
Drug-induced dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT04483583/Prot_SAP_001.pdf